CLINICAL TRIAL: NCT00457288
Title: Efficacy and Safety of TF002 in Cutaneous Mastocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JADO Technologies GmbH (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MICUMA
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-11

CONDITIONS: Cutaneous Mastocytosis
Keywords: Cutaneous Mastocytosis; Topical treatment
MeSH Terms: conditions — Mastocytosis, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: TF 002

SUMMARY:
The current study will investigate the effects of TF002 on cutaneous mastocytosis or cutaneous involvement of systemic mastocytosis as compared to clobetasol proprionate (positive control) and a general skin care product without active ingredient targeting mastocytosis (negative control) based on clinical effects on Darier´s signs and the histological evaluation of mast cell numbers in skin bioptic material.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo- and active-controlled study with intra-individual comparison of test areas.

The primary study target is to evaluate the safety and efficacy of TF002 for the treatment of cutaneous mastocytosis or systemic mastocytosis with skin involvment. The treatment period of 14 days was adjusted to the maximum recommended treatment period for the comparator Dermoxinale®.

Since there are no approved therapies for this indication a placebo controlled design was chosen.

There are some reports about transient treatment effects using high potent steroids like clobetasol in mastocytosis. This triggered the decision to use Dermoxinale® as positive control.

To validate the clinical scores used in the study, surrogate markers describing the Darier´s sign (thermography, volumetric test) will be evaluated optionally.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stable symptomatic maculopapulous cutaneous mastocytosis or systemic mastocytosis with involvement of the skin and with positive Darier's Sign
* 3 comparable skin lesional areas
* Otherwise healthy according to physical examination
* Informed consent signed and dated

Exclusion Criteria:

* Aggressive systemic mastocytosis
* Other dermatological diseases at treated skin site
* Known hypersensitivity to study drugs or their components
* Mental disorders
* Drug or alcohol dependency
* Any other chronic or acute illness requiring systemic treatment which might have any influence on the outcome of the study in the 4 weeks before start of treatment and during the study (investigator's decision).
* Immunodeficiency including HIV
* Pregnancy or lactation
* Participation in another clinical trial within the last 30 days
* Malignant skin lesions
* Radiation therapy of target areas excluding UV therapy longer then 4 weeks before start of study treatment
* Dermal comorbidities within the target areas
* Any concomitant medication which might influence the study objectives or are known to provoke or aggravate mastocytosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of treatment response

SECONDARY OUTCOMES:
Number of skin mast cells
Volumetric and thermographic analyses

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, Prof, Principal Investigator — Charite University, Berlin, Germany
Locations (4):
- Germany (4):
  - Klinik und Poliklinik für Dermatologie und Venerologie der Universität, Cologne, Köln
  - Universitäts-Hautklinik, Mainz
  - Klinik und Poliklinik für Dermatologie und Allergologie der LMU, München
  - Klinik und Poliklinik für Dermatologie und Allergologie am Biederstein der TU, München